CLINICAL TRIAL: NCT06194643
Title: Pregnancy Outcomes and Platelet PhenotYpes (POPPY)
Brief Title: Platelets in Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22-01439
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood RNA and DNA will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant people at high risk of preeclampsia (case group): Investigators will collect a sample of blood (up to 50ml) at the time of a previously scheduled visit as part of routine prenatal care. Platelet phenotyping, measuring platelet activity, and the platelet transcriptome will be performed on samples. Plasma, serum, whole blood RNA and DNA will be collected.
- Pregnant people at low risk of preeclampsia (control group): Investigators will collect a sample of blood (up to 50ml) at the time of a previously scheduled visit as part of routine prenatal care. Platelet phenotyping, measuring platelet activity, and the platelet transcriptome will be performed on samples. Plasma, serum, whole blood RNA and DNA will be collected.

SUMMARY:
This is a prospective observational cohort study of platelet phenotype in pregnant patients at high-risk for the development preeclampsia. Blood samples will be collected prior to the initiation of daily aspirin and again in the second trimester to evaluate for platelet changes during pregnancy in patient's as a result of aspirin use and their association with adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria (Case Group):

* Pregnant patients receiving prenatal care prior to 17 weeks at NYU Langone Health- Obstetrics & Gynecology Associates
* Age 18-50 years
* Singleton viable gestation
* Pregnant patients at high risk of preeclampsia: Patients meeting USPSTF recommendation for low-dose aspirin (81 mg/day) prophylaxis for preeclampsia based on clinical risk factors (see below)

Inclusion Criteria (Control Group):

* Pregnant patients receiving prenatal care prior to 17 weeks at NYU Langone Health- Obstetrics & Gynecology Associates
* Age 18-50 years
* Singleton viable gestation
* Pregnant patients at low risk of preeclampsia: Patients who do not meet USPSTF recommendation for low-dose aspirin (81 mg/day) prophylaxis for preeclampsia based on clinical risk factors.

Exclusion Criteria (Case and Control Group):

* Allergy to aspirin
* Antithrombotic or antiplatelet therapy
* Anemia (hemoglobin <10 g/dl) or thrombocytopenia (Platelet count <100,000), or thrombocytosis (Platelet count >600)
* Known hemorrhagic diathesis
* Planned delivery outside of NYU

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant people at high and low risk of preeclampsia and other adverse perinatal outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Individuals with Overactive Platelets | Blood Draw 1 (taken between Weeks 6 and 14)
Number of Individuals with Overactive Platelets | Blood Draw 2 (taken between Weeks 24 and 28)

SECONDARY OUTCOMES:
Incidence of Adverse Pregnancy Outcomes | Day 30 Post-Delivery (Up to Month 11)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A. Penfield, MD, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the primary results reported in this article, after deidentification (text, tables, figures, and appendices), will be shared with investigators who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Data sharing will begin 9 months and end 36 months following article publication or as required by a condition of awards and agreements supporting the research. Requestors must execute a data use agreement with NYU Langone Health. Requests may be directed to: christina.penfield@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Data will be shared with investigators who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Requests should be directed to christina.penfield@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.